CLINICAL TRIAL: NCT03823118
Title: S1 Plus Anlotinib in Treating Patients With Refractory or Relapsed Small-cell Lung Cancer：An One-arm, Phase Ⅱ, Multi-center Clinical Study (SALTER TRIAL)
Brief Title: S1 Plus Anlotinib in Treating Patients With Refractory or Relapsed Small-cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Head of Department of Radiation Oncology, Taizhou Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALTER Trial
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Small Cell Lung Cancer Recurrent

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S1/Anlotinib (Experimental): Anlotinib 12mg qd, day 1 to day 14 followed by 7 days off treatment in a 21-day cycle until maximum 6 cycles； S1 60mg bid, day 1 to day 14 followed by 7 days off treatment in a 21-day cycle until it can not tolerate, or disease progression.
  Interventions: Drug: S1/Anlotinib

INTERVENTIONS:
Drug: S1/Anlotinib — Anlotinib 12mg qd, day 1 to day 14 followed by 7 days off treatment in a 21-day cycle until maximum 6 cycles； S1 60mg bid, day 1 to day 14 followed by 7 days off treatment in a 21-day cycle until it can not tolerate, or disease progression.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of S1 combination with Anlotinib in patients with small cell lung cancer whose cancer has progression or recurrence after at least one standard chemotherapy.

DETAILED DESCRIPTION:
Although SCLC is very responsive to initial treatment, most patients relapse with relatively resistant disease.These patients have a median survival of only 4 to 5 months when treated with further systemic therapy. Improvements in therapy for relapsed SCLC are much needed.The purpose of this study is to assess the efficacy and safety of S1 combination with Anlotinib in patients with small cell lung cancer whose cancer has progression or recurrence after at least one standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologically confirmed small cell lung cancer;
* Systemic chemotherapy that has previously received at least one or more lines regimen, followed by disease progression or recurrence;
* Age 18-75 years,ECOG PS:0-2,Life expectancy of more than 3 months
* participants had at least one measurable target lesion by RECIST1.1
* The main organ function meets the following criteria:absolute value of neutrophils ≥ 1.5 × 109 / L, platelets ≥80 × 109 / L, hemoglobin ≥ 80 g / L;total bilirubin ≤ 1.5 times the upper limit of normal value, aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal value (if liver metastasis, ≤ upper limit of normal value 5 times), serum creatinine ≤ 1.5 times the upper limit of normal;
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients who have been used anti-angiogenesis inhibitors,such as (such as sunitinib,bevacizumab,endostar et al.
* Subjects with symptomatic brain metastases;
* Patients whose primary lesion with active bleeding within 4 months
* Hypertension, which is uncontrolled by the drug, is defined as: systolic blood pressure ≥ 160 mmHg, or diastolic blood pressure ≥ 100 mmHg
* Patients with active or unable to control serious infections
* Patients who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | each 21 days up to the toxicity or PD (up to 6 months)
  measured by Response Evaluation Criteria in Solid Tumors version 1.1
progression-free survival (PFS) | Duration of time from the start of treatment to the first documented disease progression according to RECIST 1.1 or death due to any cause, whichever occurs first, assessed up to 12 months
  PFS will be estimated using standard Kaplan Meier survival analysis methods.

SECONDARY OUTCOMES:
Overall survival (OS) | Duration of time from the start of treatment to date of death, assessed up to 2 years
  OS will be estimated using standard Kaplan Meier survival analysis methods.
Incidence of adverse events | Up to 2 years
  Incidence of adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Taizhou Hospital, Wenzhou Medical University, Taizhou, Zhejiang
  - Enze Hospital, Taizhou, Zhejiang
  - Sanmen People's Hospital, Taizhou, Zhejiang

REFERENCES:
- [Derived] Wang W, Wu G, Luo W, Lin L, Zhou C, Yao G, Chen M, Wu X, Chen Z, Ye J, Yang H, Lv D. Anlotinib plus oral fluoropyrimidine S-1 in refractory or relapsed small-cell lung cancer (SALTER TRIAL): a multicenter, single-arm, phase II trial. BMC Cancer. 2024 Sep 27;24(1):1182. doi: 10.1186/s12885-024-12954-8. PMID 39333988